CLINICAL TRIAL: NCT05316883
Title: Biomarkers in Clozapine-responding Schizophrenia
Acronym: BiCS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jimmi Nielsen (Other)
Responsible Party: Sponsor-Investigator, Jimmi Nielsen, Professor, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BiCS2019
Record Dates: First submitted 2020-09-30; First posted 2022-04-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Clozapine

STUDY DESIGN:
Intervention Model Description: To compare biomarkers between clozapine responders and non-responder before and after 12 weeks of treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- clozapine treatment (Other): Open label clozapine will be given to all participants in clinical doses adjusted to sideeffects and clinical effect
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Clozapine — clinical doses adjusted to sideeffects and clinical effect

SUMMARY:
The outline of the current project is to establish a cohort of patients with treatment refractory schizophrenia eligible for clozapine, to identify clinical and biological characteristics of clozapine responding patients. Patients will be offered treatment with clozapine according to national clinical guidelines. Before clozapine is initiated, patients will be offered a thoroughly neurobiological examination, and re-examination will be carried out after 12 weeks of treatment. The primary focus of the examinations will be immunological markers and autoantibodies in the blood and cerebrospinal fluid, permeability of the blood-brain barrier and magnetic resonance imaging of structural, neurochemical and functional brain changes.

DETAILED DESCRIPTION:
Patients will be examined before and after 12 weeks of treatment with clozapine

Examinations at baseline and follow up will be:

* Clinical ratings
* Blood inflammatory markers
* Inflammatory markers in cerebro spinal fluid
* MRI : examination of grey & white matter, glutamate and GABA in Anterior Cingulate cortex and glutamate in thalamus,
* selected cognitive measures

ELIGIBILITY:
Inclusion Criteria:

* According to ICD-10 fulfill diagnostic criteria for schizophrenia (F20.x), chronical paranoid psychoses (F22), Schizoaffective psychoses (F25) or other non-organic psychoses (F28/F29);
* Age 18-65 years;
* Legally competent;
* Stabil antipsychotic treatment during last month
* Being treatment refractory according to TRIPP-guidelines (Howes et al. 2017) defined as having tried at least two antipsychotic drugs in sufficient dosage (≥600 mg chlorpromazine equivalent) for a sufficient time (≥ 6 weeks) without sufficient symptom improvement (still a moderate level of positive symptoms).
* Recreational use of substances is allowed as long as it does not interfere with compliance
* Fertile females must use safe contraception (spiral or any hormonal contraception).

Exclusion Criteria:

* Involuntarily psychiatric admittance during the study
* Substance abuse that interfere with compliance
* Pregnancy (will be verified by urine-HCG-test in fertile females)
* Toxic or idiosyncratic agranulocytosis in the past
* Reduced bone marrow function according to blood samples
* According to information from patient and available files, noUncontrolled

  * Current uncontrolled epilepsy
  * Current circulatory collapse and / or CNS depression for any cause
  * Current severe kidney, heart or liver disease
  * Current paralytic ileus

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-02-28 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Qalb | Baseline
  Quotient albumin (Qabl) in cerebrospinal fluid (CSF) compared to plasma
Change in Qalb | Baseline and after 12 weeks
  Change in quotient albumin in cerebrospinal fluid compared to plasma
Change in IL-6 and TGF-beta | Baseline and after 12 weeks
  Change in interleukin 6 (IL-6) and transcription growth factor beta (TGF-beta)

SECONDARY OUTCOMES:
Change in FA, MD, AD and RD | Baseline and after 12 weeks
  Change in fractional anisotropy (FA), mean diffusivity (MD), axial diffusivity (AD) and radial diffusivity (RD)
Change in cortical thickness as measured with FreeSurfer | Baseline and after 12 weeks
  Change in cortical thickness as measured with FreeSurfer
Change in glutamate in ACC and thalamus measured with MTI | Baseline and after 12 weeks
  Change in glutamate in anterior cingulate cortex (ACC) and thalamus measured with magnetic transfer imaging (MTI)

CONTACTS AND LOCATIONS:
Overall Officials: Jimmi Nielsen, PhD, Principal Investigator — Mental health Service, Glostrup
Locations (1):
- Mental Health Services Glostrup, Unit for Complicated Schizophrenia, Glostrup Municipality, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No